CLINICAL TRIAL: NCT02292940
Title: Consumer Health IT Tools: Impact on Patient Experience, Access, and Health Outcomes for Patients With Complex Chronic Conditions
Brief Title: Consumer Health IT Tools: Impact on Experience, Access, and Outcomes for Patients With Complex Chronic Conditions
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CN-13-1567-H
Record Dates: First submitted 2014-10-30; First posted 2014-11-18 (Estimated); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Chronic Disease; Patient Outcome Assessment; Electronic Health Records
Keywords: patient outcome assessment; electronic health records
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patient use of health IT tools to interact with healthcare providers and delivery systems, including exchanging secure messages with their medical providers and using other web-based tools, has great potential to increase patient access to care, change the way healthcare is delivered, and affect patient clinical outcomes. This study will examine the impact of implementation and use of consumer health IT tools on patient-reported access to care, utilization of medical care services, and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic conditions
* Patient had at least 10-month membership in 2005

Exclusion Criteria:

* Patients less than age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a chronic disease
Sampling Method: Non-Probability Sample
Enrollment: 168477 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Reed, DrPh, Principal Investigator — Kaiser Permanente

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients with at least 10-month membership in 2005
Pre-assignment Details: Note: the participants in the Medical Record only arm of the study and the participants in the Survey arm of the study are two different groups of participants. The Medical Record arm of the study includes data from January 2006 to December 2007. The Survey was completed between March 2015 and April 2016.
Groups:
- Adult Patients With Chronic Conditions: Medical Record Data: Medical record data of adult patients with diabetes and/or complex chronic conditions in a large integrated delivery system.
- Adult Patients With Chronic Conditions: Survey Data: Survey data completed by adult patients with diabetes and/or complex chronic conditions in a large integrated delivery system. Participants were given the option to complete the survey by mail, by phone with a research assistant, or online.
Period: Overall Study
Arm/Group | Adult Patients With Chronic Conditions: Medical Record Data | Adult Patients With Chronic Conditions: Survey Data
Started | 165477 | 3000
Completed | 165477 | 1824
Not Completed | 0 | 1176

BASELINE CHARACTERISTICS:
Groups:
- Adult Patients With Chronic Conditions Survey Data: Survey data competed by adult patients with diabetes and/or complex chronic conditions in a large integrated delivery system. Participants were given the option to complete the survey by mail, by phone with a research assistant, or online
- Total: Total of all reporting groups
Arm/Group | Adult Patients With Chronic Conditions: Medical Record Data | Adult Patients With Chronic Conditions Survey Data | Total
Number analyzed (Participants) | 165,477 | 1824 | 167301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 92,005 | 941 | 92946
  >=65 years | 73,472 | 883 | 74355
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79,594 | 948 | 80542
  Male | 85,883 | 876 | 86759
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 165,477 | 1824 | 167301

OUTCOME MEASURES:

1. Primary Outcome: Number of Ambulatory Care Sensitive Conditions (ACSC) Hospitalizations. Portal Users vs Those Who Are Not Portal Users
Description: Number of ambulatory care sensitive conditions (ACSC) hospitalizations per 1000 patients per month among those who accessed the portal and those who did not access the portal.
Time Frame: Data from 2006-2007
Population: Only those participants who had an event (ACSC Hospitalization) were included in this analysis.
Measure: Number; unit: hospitalizations/1000 participants/month
Groups:
- ACSC Hospitalizations for Those Accessing the Portal: ACSC Hospitalizations for those accessing the portal.
- ACSC Hospitalizations - Non Portal Users.: ACSC Hospitalizations for those who did not access the portal.
Arm/Group | ACSC Hospitalizations for Those Accessing the Portal | ACSC Hospitalizations - Non Portal Users.
Number analyzed (Participants) | 36,983 | 128,494
hospitalizations/1000 participants/month | 6.2 | 7.0

2. Primary Outcome: Patient Self-report Survey Data
Description: Patient-reported reasons for using the patient portal
Time Frame: March 2015-April 2016
Population: Only those participants completing a survey and indicating that they used the portal were included in this analysis.
Measure: Number; unit: participants
Groups:
- Survey Data: Portal Users: Adult patients with complex chronic conditions who registered to use the portal completed a survey describing reasons for using the portal.
Arm/Group | Survey Data: Portal Users
Number analyzed (Participants) | 1392
participants
  Use portal because it is convenient | 1252
  Use portal to access data/information | 1284
  Say the portal integrates with other health care | 1285

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected/assessed are therefore all are recorded as 0
Description: Adverse Events were not collected/assessed and therefore all are recorded as 0
Groups:
- Adult Patients With Complex Chronic Conditions: Adult patients with diabetes and/or complex chronic conditions in a large integrated delivery system.
- Adult Patients With Complex Chronic Conditions: Survey Data: Survey data completed by adult patients with diabetes and/or complex chronic conditions in a large integrated delivery system. Participants were given the option to complete the survey by mail, by phone with a research assistant or online.
Arm/Group | Adult Patients With Complex Chronic Conditions | Adult Patients With Complex Chronic Conditions: Survey Data
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No